CLINICAL TRIAL: NCT02965027
Title: Prazosin for the Prophylaxis of Chronic Post-Traumatic Headaches in OEF/OIF/OND Service Members and Veterans With Mild TBI
Brief Title: Prazosin for Post-Concussive Headaches
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency); Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W81XWH-15-2-0060
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Post-Traumatic Headache
Keywords: Chronic Headache; Post-Traumatic Stress Disorder; Iraq/Afghanistan Veteran
MeSH Terms: conditions — Post-Traumatic Headache; Headache Disorders; Stress Disorders, Post-Traumatic | interventions — Prazosin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prazosin (Experimental): Prazosin capsules beginning at 1 mg orally at bedtime. Titrate over 5 weeks to maximum dose of 5 mg in the morning and 20 mg at bedtime.
  Interventions: Drug: Prazosin
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prazosin
  Other Names: Minipress
  Arms: Prazosin
Drug: Placebo
  Other Names: inactive substance, sugar pill
  Arms: Placebo

SUMMARY:
Mild traumatic brain injury (mTBI) caused by blast effects of explosive devices has been called the "signature injury" of soldiers who served in the Iraq and Afghanistan conflicts. mTBI can also occur from impact or hitting the head on an object or the ground. Although termed "mild" in comparison to major brain injuries, people with mTBI can have problems with their memory and concentration. People with mTBI can also find they are more irritable, have more anxiety, and have trouble with their mood and sleep.

The purpose of this study is to see if a medication called prazosin can help treat chronic headaches in people with mTBI. The Food and Drug Administration (FDA) has approved prazosin for treating people with high blood pressure. At this time, the FDA has not approved prazosin in the treatment of mTBI or headaches. Some people who have posttraumatic stress disorder (PTSD) and have been taking prazosin for their medical conditions or who have taken it in research studies have said they have fewer headaches.

DETAILED DESCRIPTION:
Background and Rationale: Headaches following mild traumatic brain injury (mTBI) are common, can be refractory to standard therapies, and may persist and worsen to become a debilitating chronic pain syndrome. The purpose of this study is to evaluate the centrally acting alpha-1 adrenoreceptor (AR) antagonist drug prazosin as a prophylactic treatment for chronic posttraumatic headaches (PTHAs). The impetus for this study comes from a large open-label case series in Iraq and Afghanistan Veterans with mTBI and PTHAs and data from a placebo-controlled trial evaluating use of prazosin for posttraumatic stress disorder (PTSD) in active-duty Servicemembers (SMs). Findings from these studies showed that in addition to decreasing PTSD-related symptoms and improving sleep quality, prazosin decreased the frequency and severity of headaches, which were common in the study populations.

Study Objectives, Specific Aims, and Hypotheses: The objective of this study is to evaluate the efficacy of prazosin as a prophylactic treatment for persistent PTHAs, which will be accomplished by conducting a randomized placebo-controlled double blind trial of prazosin vs. placebo in active-duty SMs and Veterans who were in military service at any time from October 7, 2001 to the present with persistent PTHAs.

* Specific Aim 1: To determine the effect of prazosin compared to placebo on headache frequency, headache severity and duration, use of abortive/analgesic medications, and headache-related disability.
* Specific Aim 2: To determine the effect of prazosin on sleep disturbance, PTSD symptoms, depressive symptoms, alcohol consumption, global cognitive function, health-related quality of life, and global clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Active-duty Servicemembers (SMs) or Veterans aged 18 or older who are in good general health.
* History of blast and/or impact head trauma mild traumatic brain injury (mTBI) meeting Defense and Veterans Brain Injury Center (DVBIC) mTBI criteria.

  o Mild TBI is defined as an injury to the head causing at least one of the following: alteration in consciousness (for up to 24 hours after the injury), loss of consciousness (0-30 minutes), and/or post-traumatic amnesia (up to 1 day post-injury). If available, the Glasgow Coma Scale score must be 13-15, and head imaging findings (if imaging was performed) must be negative.
* Frequent headaches (HAs) that started within 3 months after a head injury or marked worsening (a two-fold or greater increase in frequency and/or severity) of pre-existing headaches within 3 months of head injury.

  * HAs either 1) must last 4 or more hours a day and reach a moderate to severe intensity at any point during the headache, or 2) may be of any severity or duration if the participant takes a medication or other agent in an effort to stop or treat a headache.
  * HAs meeting these criteria must have been present on average at least 8 days per 4-week period and occurring at a stable level by self-report for at least 3 months prior to the Initial Screening Visit. The 4-week HA frequency/severity criteria must be confirmed during the Preliminary Screening Period.
* Participants of childbearing potential must agree to abstain from sexual relations that could result in pregnancy or use an effective method of birth control acceptable to both participant and the clinician prescriber during the study. Participants who are not of childbearing potential are not required to use contraception during the study.
* Participants must have English fluency sufficient to complete study measures.

Exclusion Criteria:

* Participation in other interventional research.
* History of penetrating head injury
* History of TBI more severe than mild by DVBIC criteria
* A primary non migraine and/or tension-type HA disorder (for example hemicrania continua; cluster) that accounts for the majority of current symptoms.
* HAs of any kind of moderate or severe intensity on an average of more than 4 days per month preceding the concussive trauma
* Acute or serious medical illness or unstable chronic medical illness (e.g., unstable angina, myocardial infarction within 6 months, congestive heart failure, clinically significant or concerning cardiac arrhythmias; preexisting hypotension [systolic blood pressure<110] or orthostatic hypotension [systolic drop >20 mm Hg after 2 min standing accompanied by lightheadedness], chronic renal or hepatic failure, or acute pancreatitis. The eligibility of potential participants having acute serious and/or chronic medical illnesses other than those listed will be evaluated on a case-by-case basis by a study physician, physician assistant - certified (PA-C), or advanced registered nurse practitioner (ARNP).
* Use of prazosin or other alpha-1 antagonist (including but not limited to alfuzosin, doxazosin, silodosin, tamsulosin, terazosin) for any purpose in the 2 weeks prior to initial screen (P1) visit and prohibited throughout the study
* Allergy or previous adverse reaction to prazosin or other alpha-1 antagonist
* Active psychosis or psychotic disorder, severe depression (as determined per clinician prescriber judgment), severe psychiatric instability or severe situational life crisis (including evidence of being actively suicidal or homicidal).
* Meets Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for any Substance Use Disorder except caffeine-related disorders, or tobacco-related disorders.
* History of delirium within the prior 3 months, epilepsy, stroke, dementia, psychotic disorder, or bipolar disorder
* Structural brain abnormalities on any prior imaging with associated clinically evident manifestations
* Current participation in transcranial magnetic stimulation studies
* Women of childbearing potential must not be pregnant, planning to become pregnant during the study period, or nursing.
* Participation in a HA support group or other activity such as meditation or yoga intended to mitigate HA or other chronic pain must be stable at least 4 weeks prior to beginning the initial screen (P1) visit and may not be started during the study
* Failure to record HA data for at least 80% of days during the Screening Period
* Not suitable for study per clinician judgement.

Medication-and other Treatment-Related Considerations:

* The use of HA rescue or symptom-relieving medications will be allowed during the study. This includes triptans, ergotamines, opioids, simple analgesics (e.g. acetaminophen, aspirin, or non-steroidal anti-inflammatories [NSAIDS], and combination analgesics. Their use will be recorded on the concurrent medication case report form (CRF) during the Preliminary Screening Period (P1) and throughout the remainder of the study. Randomization of participants will be stratified based on whether their use of HA medications meets International Classification of Headache Disorders 3rd addition (ICHD-3 beta) criteria for overuse of these medications, as described in section 5.5 below.
* Opioid Medications: Use of opioids for treatment of HA or non-HA-related pain or for any other purpose is allowed during the study. Any opioid use would ideally be excluded due to potential confounding effects on interpretation of response to treatment. However, in this population, particularly in Veterans with chronic pain or undergoing minor orthopedic or dental procedures, opioid use is common. Use of opioids, including frequency and dose, will be recorded on the concurrent medication CRF.
* Cannabis: The use of cannabis in any form is not excluded unless its use meets criteria for Cannabis Use Disorder. All use of cannabis will be documented.
* Other Medications: Participants who are using other medications or treatments on a routine basis must be on a stable dose for at least 4 weeks prior to the Preliminary Screening Period (P1), and must intend to continue the medication at the same regimen for the duration of the trial unless lack of efficacy, safety, or tolerability dictates otherwise. The following medications and treatments are not excluded:

  * Psychoactive drugs (for example, anticonvulsants, benzodiazepines, antidepressants, sedative/hypnotics),
  * Antihypertensive medications (including beta-blockers, calcium channel blockers, angiotensin converting enzyme [ACE] inhibitors, and angiotensin receptor blockers),
  * The use of magnesium in any dose that is prescribed for the purpose of HA prevention or treatment. The incidental use of magnesium in multi-vitamins, laxatives, etc. is permissible but must be documented.
  * Hormones (for example, testosterone, estrogen, or progesterone) in any form.
  * Onabotulinum toxin A and nerve block injections for the purpose of HA prevention are permissible if the treatment response has been stable during the two most recent treatment cycles.
  * The "as-needed" (prn) use of any non-exclusionary medications is allowed; however, such use must be discussed with a clinician prescriber and documented.
* The use of butalbital in any form within 4 weeks of beginning the Preliminary Screening Period (P1) through the end of the participant's study involvement is exclusionary.
* Participants who have been taking trazodone will undergo a 2-week washout period before the Preliminary Screening Period (P1 visit). Combining prazosin and trazodone may increase the risk of priapism. We have decided to begin the washout period before the Preliminary Screening Period in order to remove any confounding variables while on the headache log and actigraphy.
* Sildenafil (Viagra), tadalafil (Cialis), vardenafil (Levitra), and avanafil (Stendra) will not be permitted during the study drug dose Titration Period, because of increased risk of hypotension in combination with alpha-1 blockers, but will be allowed at half the usual starting dose following the study drug dose Titration Period, per VA prescribing guidelines.
* Use of supplements containing nitrates and supplements containing stimulants (such as ephedra) are exclusionary in the two weeks prior to initial screen (P1) visit and prohibited throughout the study. Participants who take these supplements will be asked to discontinue them for a minimum of two weeks before the Preliminary Screening Period (P1 visit).
* Use of prescribed stimulants (such as amphetamine or dextroamphetamine containing medications) is exclusionary in the 2 weeks prior to the initial screen (P1) visit and prohibited throughout the study. Participants who take these medications will be asked to discontinue them for a minimum of 2 weeks before the Preliminary Screening Period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray A Raskind, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (2):
- United States (2):
  - VA Puget Sound Health Care System, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Prazosin: Prazosin capsules beginning at 1 mg orally at bedtime. Titrate over 5 weeks to maximum dose of 5 mg in the morning and 20 mg at bedtime.
  Prazosin
- Placebo: Placebo capsules
  Placebo
Period: Overall Study
Arm/Group | Prazosin | Placebo
Started | 59 | 30
Completed | 52 | 26
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin | Placebo | Total
Number analyzed (Participants) | 59 | 30 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 57 | 30 | 87
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (11.9) | 37.6 (10.1) | 38.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 53 | 25 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 5 | 16
  Not Hispanic or Latino | 34 | 20 | 54
  Unknown or Not Reported | 14 | 5 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 2 | 0 | 2
  Asian | 2 | 1 | 3
  Black | 12 | 8 | 20
  White | 31 | 18 | 49
  Hawaiian Native or Pacific Islander | 2 | 0 | 2
  Missing/Unknown | 3 | 0 | 3
  More than one race | 5 | 0 | 5
  Other | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 59 | 30 | 89

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Headache Frequency
Description: Headache log completed by participant to capture number of headaches experienced.
Time Frame: baseline, 4,8, and 12 weeks after steady dose
Measure: Mean (Standard Error); unit: headaches per month
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 59 | 30
headaches per month
  Baseline | 16.4 (1.2) | 18.5 (1.6)
  Week 4 - Baseline | -9.2 (0.9) | -7.4 (1.2)
  Week 8 - Baseline | -9.9 (0.9) | -9.1 (1.2)
  Week 12 - Baseline | -10.7 (0.9) | -6.9 (1.3)

2. Secondary Outcome: Overall Sleep Quality as Assessed by Pittsburgh Sleep Quality Index
Description: Overall sleep quality assessed utilizing the Pittsburgh Sleep Quality Index (PSQI). The PSQI contains 19 self-rated questions. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. The seven component scores are then added to yield one "global" score with a range of 0-21 points, "0" indicating no difficulty and "21" indicating sever difficulty in all areas.
  Minimum Score = 0 (better); Maximum Score = 21 (worse). Interpretation: TOTAL < 5 associated with good sleep quality. TOTAL > 5 associated with poor sleep quality The difference between means is shown for weeks 4, 8 and 12.
Time Frame: baseline, 4, 8, 12 weeks after steady dose
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 59 | 30
score on a scale
  Baseline | 12.1 (0.6) | 12.0 (0.8)
  Week 4 - Baseline | -1.0 (0.5) | 0.1 (0.7)
  Week 8 - Baseline | -1.9 (0.5) | -0.9 (0.7)
  Week 12 - Baseline | -2.2 (0.5) | -0.8 (0.7)

3. Secondary Outcome: Insomnia Severity Index
Description: Insomnia severity assessed using the Insomnia Severity Index (ISI). This 7-item self-report is designed to measure and detect cases of insomnia. Each question is scored on a scale of 0 to 4. The 7 items are added together.
  Sum scores for items 1-7 0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe) The difference between means is shown for weeks 4, 8 and 12.
Time Frame: baseline, 4, 8, 12 weeks after steady dose
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 59 | 30
score on a scale
  Baseline | 16.9 (0.8) | 17.6 (1.2)
  Week 4 - Baseline | -3.3 (0.7) | -0.5 (1.0)
  Week 8 - Baseline | -3.1 (0.7) | -1.0 (1.0)
  Week 12 - Baseline | -3.7 (0.7) | -0.9 (1.0)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Prazosin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/59 | 1/30
Other Adverse Events (participants affected / at risk) | 52/59 | 22/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin (N=59) | Placebo (N=30)
planned surgical procedure (Surgical and medical procedures) | 1 (1) | 0 (0) — anterior cervical discectomy and fusion
planned surgical procedure (Surgical and medical procedures) | 0 (0) | 1 (1) — nasal endoscopy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin (N=59) | Placebo (N=30)
Dizziness (any) (General disorders) | 37 (51) | 6 (7)
Dizziness on Standing (General disorders) | 24 (30) | 1 (1)
Lightheadedness (General disorders) | 28 (32) | 11 (11)
Vertigo (General disorders) | 1 (1) | 1 (1)
Nasal Congestion (General disorders) | 19 (21) | 3 (3)
Headache worsening (General disorders) | 2 (2) | 4 (5)
Drowsiness/Lethargy (General disorders) | 26 (30) | 5 (5)
Low Energy (General disorders) | 16 (17) | 3 (3)
Weakness (generalized) (General disorders) | 6 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 20 (25) | 4 (4)
Palpitations (Cardiac disorders) | 21 (23) | 6 (6)
Incontinence (Renal and urinary disorders) | 4 (4) | 0 (0)
Peripheral Edema (General disorders) | 11 (12) | 3 (4)
Insomnia (General disorders) | 8 (10) | 2 (2)
Depression or depressed mood (Psychiatric disorders) | 7 (7) | 2 (2)
Suicidal Ideation (Psychiatric disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT02965027/Prot_SAP_000.pdf